CLINICAL TRIAL: NCT03783507
Title: Foods Within a Meal and Food Liking Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Tennessee, Knoxville (Other)
Responsible Party: Principal Investigator, Hollie Raynor, Associate Dean of Research, The University of Tennessee, Knoxville
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Screening
Other Study IDs: UTK IRB-18-04832-XP
Record Dates: First submitted 2018-12-02; First posted 2018-12-21 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Diet Habit; Obesity
Keywords: Energy Density
MeSH Terms: conditions — Feeding Behavior; Obesity

STUDY DESIGN:
Intervention Model Description: In order to examine if low-ED foods and high-ED foods substitute for each other, a 4 X 4 mixed-factor design with a between-subjects factor of order and a within-subjects factor of meal will be used. For the within-subjects factor of meal, four meal conditions will be implemented. Participants will be randomized to one of 4 orders to reduce the possibility of an order effect. During all sessions, participants will be provided with 12 ounces of water.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Order 1 (Experimental): Meal 1, Meal 2, Meal 3, Meal 4
  Interventions: Behavioral: Order 1
- Order 2 (Experimental): Meal 2, Meal 3, Meal 4, Meal 1
  Interventions: Behavioral: Order 2
- Order 3 (Experimental): Meal 3, Meal 4, Meal 1, Meal 2
  Interventions: Behavioral: Order 3
- Order 4 (Experimental): Meal 4, Meal 1, Meal 2, Meal 3
  Interventions: Behavioral: Order 4

INTERVENTIONS:
Behavioral: Order 1 — Meal Order 1:
  Meal Session 1 participant receives meal 1 (3 low-ED, 0 medium-ED, 2 high-ED) Meal Session 2 participant receives meal 2 (3 low-ED, 1 medium-ED,1 high-ED) Meal Session 3 participant receives meal 3 (1 low-ED, 2-medium ED, 2 high-ED) Meal Session 4 participant receives meal 4 (1 low-ED, 3 medium-ED, 1 high-ED)
  Arms: Order 1
Behavioral: Order 2 — Meal Order 2:
  Meal Session 1 participant receives meal 2 (3 low-ED, 1 medium-ED,1 high-ED) Meal Session 2 participant receives meal 3 (1 low-ED, 2-medium ED, 2 high-ED) Meal Session 3 participant receives meal 4 (1 low-ED, 3 medium-ED, 1 high-ED) Meal Session 4 participant receives meal 1 (3 low-ED, 0 medium-ED, 2 high-ED)
  Arms: Order 2
Behavioral: Order 3 — Meal Order 3:
  Meal Session 1 participant receives meal 3 (1 low-ED, 2-medium ED, 2 high-ED) Meal Session 2 participant receives meal 4 (1 low-ED, 3 medium-ED, 1 high-ED) Meal Session 3 participant receives meal 1 (3 low-ED, 0 medium-ED, 2 high-ED) Meal Session 4 participant receives meal 2 (3 low-ED, 1 medium-ED,1 high-ED)
  Arms: Order 3
Behavioral: Order 4 — Meal Order 4:
  Meal Session 1 participant receives meal 4 (1 low-ED, 3 medium-ED, 1 high-ED) Meal Session 2 participant receives meal 1 (3 low-ED, 0 medium-ED, 2 high-ED) Meal Session 3 participant receives meal 2 (3 low-ED, 1 medium-ED,1 high-ED) Meal Session 4 participant receives meal 3 (1 low-ED, 2-medium ED, 2 high-ED)
  Arms: Order 4

SUMMARY:
For weight loss to occur, energy intake needs to be reduced to incur an energy deficit. One dietary strategy that may facilitate weight loss is consuming a diet low in dietary energy density (ED). It is hypothesized that a diet low in ED, which can be achieved by a high intake of low-ED foods, low intake of high-ED foods, or a combination of the two, will allow a greater amount of volume of food to be consumed relative to energy consumed, which can assist with reducing energy intake.

To understand how best to lower the ED of the diet, it is important to understand the relationship between low-ED and high-ED foods. Behavioral economics is a framework that provides a foundation to understand that eating behaviors can be substitutes for each other. Substitute eating behaviors are two behaviors that change in the opposite direction of each other (i.e. one behavior increases as the other behavior decreases). If low-ED and high-ED foods are substitutes for each other, in situations in which low-ED food intake increases, high-ED food should automatically decrease, and vice versa. If they are not substitutes, when low-ED food intake increases, high-ED food intake should remain unchanged, and when high-ED food intake decreases, low-ED food intake should remain unchanged. When low-Ed and high-ED foods are not substitutes for each other, purposeful change in intake for both low- and high-ED foods need to occur to best lower dietary ED.

Thus, the purpose of this study is to investigate if low-ED foods and high-ED foods substitute for each other. Healthy weight adults will be served a meal over 4 sessions, with each meal containing 5 different food items. The foods in the meal will vary in ED: low-ED = 0 to 1.0 kcal/kg; medium-ED = 1.1 to 2.9 kcal/kg; high-ED = > 3.0 kcal/g. For the 4 sessions, the meals will include: 1) 3 low-ED foods, 0 medium-ED foods, 2 high-ED foods; 2) 3 low-ED foods, 1 medium-ED food, 1 high-ED food; 3) 1 low-ED food, 2-medium ED foods, 2 high-ED foods; and 4) 1 low-ED food, 3 medium-ED foods, and 1 high-ED food.

DETAILED DESCRIPTION:
All participants will be asked to come to HEAL for 1, 60-minute screening session and 4, 30-minute meal sessions, with no more than two meal sessions occurring per week between the hours of 11:00am and 7:00pm. For each participant, each meal session will need to occur within the same two-hr time frame (i.e., all meal sessions occurring between 11am and 1pm). During the first session interested participants will sign the consent form. After signing the consent form, eligibility will be confirmed by taking height and weight measures and confirming liking of foods, using a 100mm VAS. Participants will also be given questionnaires related to demographics. Prior to attending their meal session, participants will be asked to not change their typical eating pattern in the day prior to their session (including eating before 10 am), but to not eat within 3 hours of their session, and to not engage in physical activity for 24 hours prior to the session.

For the remaining four sessions, at the start of the session the participant will be asked to recall all foods and beverages consumed 24 hours prior to the scheduled appointment. During this recall if a participant reports consuming any foods or beverages besides water within 3 hours of the appointment, the appointment will be rescheduled. Participants will also be asked if they have participated in any physical activity 24 hours prior to their scheduled appointment. If the participant answers "yes," then the appointment will be rescheduled.

After completing hunger, fullness, and liking of foods questionnaires, participants will be presented with one of the four variations of meals. The exact brand and formulation of food products may change due to local availability. However, each participant will receive consistent products (and, thus, consistent weights of each food) across all of their meals. In other words, products may vary between participants but not within a single participant. Following the presentation of the meal, participants will be instructed to taste each food and that they will have 25 minutes to eat as much or as little as they would like of the meal provided. At the completion of 25 minutes, the lunch will be removed and the participant will be asked to complete a scale for evaluating levels of hunger, fullness, and liking of the foods. The participant will also be scheduled for a subsequent session the following week at a similar time. Upon completing all 5 sessions, participants will receive a $50 gift card.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 35 years;
* body mass index (BMI) 18.5 to 24.9 kg/m2;
* unrestrained eater (≤12 on Three Factor Eating Questionnaire (TFEQ);
* chicken or tomato soup, chocolate sugar-free pudding, grapes, blueberry yogurt, macaroni and cheese, vanilla ice cream, pretzels, and honey graham snacks (rate all items ≥ 50mm on a visual analogue scale (VAS);
* report regularly eating before 10 am; and
* can complete all sessions within 8 weeks of the screening session, will be eligible for the study.

Exclusion Criteria:

* report binge eating;
* report a medical condition that influences eating;
* report allergies to foods used in the investigation;
* currently smoke;
* report dietary restrictions;
* report taking a medication that affects appetite;
* report being pregnant or breast-feeding;
* report being an athlete in training.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2018-12-13 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Meal Session 1 Consumption | After 30 minute meal
  Energy intake will be calculated based upon grams consumed, manufacturer labels, and Nutrition Data System for Research (NDSR).
Meal Session 2 Consumption | After 30 minute meal
  Energy intake will be calculated based upon grams consumed, manufacturer labels, and Nutrition Data System for Research (NDSR).
Meal Session 3 Consumption | After 30 minute meal
  Energy intake will be calculated based upon grams consumed, manufacturer labels, and Nutrition Data System for Research (NDSR).
Meal Session 4 Consumption | After 30 minute meal
  Energy intake will be calculated based upon grams consumed, manufacturer labels, and Nutrition Data System for Research (NDSR).

CONTACTS AND LOCATIONS:
Overall Officials: Hollie Raynor, PhD, Principal Investigator — University of Tennessee
Locations (1):
- University of Tennessee, Knoxville, Knoxville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rolls BJ, Drewnowski A, Ledikwe JH. Changing the energy density of the diet as a strategy for weight management. J Am Diet Assoc. 2005 May;105(5 Suppl 1):S98-103. doi: 10.1016/j.jada.2005.02.033. PMID 15867904
- [Background] Rolls BJ. The relationship between dietary energy density and energy intake. Physiol Behav. 2009 Jul 14;97(5):609-15. doi: 10.1016/j.physbeh.2009.03.011. Epub 2009 Mar 20. PMID 19303887
- [Background] Epstein, L.H.; Saelens, B.E. Behavioral Economics of Obesity: Food Intake and Energy Expenditure. In Reframing Health Behavior Change with Behavioral Economics; Bickel, W.K., Vuchinich, R.E., Eds.; Lawrence Associate, Inc.: Mahwah, NJ, USA, 2000; pp. 293-311.
- [Background] Just, D.R.; Mancino, L.; Wansink, B. Could Behavioral Economics Help Improve Diet Quality for Nutrition Assistance Program Participants? Economic Research Report No. ERR-43; U.S. Department of Agriculture: Washington, DC, USA, 2007.
- [Background] Madden, G.J. A Behavioral Economics Primer. In Reframing Health Behavior Change with Behavioral Economics; Bickel, W.K., Vuchinich, R.E., Eds.; Lawrence Associate, Inc.: Mahwah, NJ, USA, 2000; pp. 3-26.

DOCUMENTS (1):
  • Informed Consent Form (2023-11-06): https://cdn.clinicaltrials.gov/large-docs/07/NCT03783507/ICF_003.pdf